CLINICAL TRIAL: NCT00952510
Title: MaNeS (Maastricht Neck Study): Development of Chronic Disability in Neck Pain Patients After a Motor Vehicle Accident
Brief Title: Maastricht Neck Study: Cervical Range of Motion in Whiplash Patients
Acronym: MaNeS
Status: Terminated | Type: Observational
Why Stopped: Respond was to low.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: J Patijn MD PhD, Maastricht University Medical Center
Other Study IDs: MEC 09-2-069
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Whiplash Injuries
Keywords: Range of motion, articular; Cervical spine
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Whiplash patients: The cohort is based on 100 whiplash patients which underwent the measure procedure to obtain cervical range of motion.

SUMMARY:
Rationale: Neck complaints are often caused by motor vehicle accidents and particular after rear-end collision. Patients complain about neck pain after a whiplash trauma, which lead to mobility restrictions of the cervical spine. It is estimated that 20% develop a chronic pain disorder after 1 year, called a chronic whiplash syndrome.

Objective: the primary objective is to investigate the natural course of active-and passive range of motion and principally the difference score between active-and passive cervical range of motion after a whiplash trauma. The secondary objectives are: investigate the predictive value of active-and passive range of motion and chronicity. Further, the correlation between the degree of restriction of the active and passive backward flexion and chronicity will be investigated. Finally, the correlation between the possible predictive factors such as pain, ideas and feeling about pain, memory and attention, events of the last year and complaints after the motor vehicle accident and chronicity are examined.

Study design and study population: a prospective cohort of 100 whiplash patients which underwent a measurement of the cervical movements and gave permission to recontact them for further research.

ELIGIBILITY:
Inclusion Criteria:

* Patients have had a measurement of the cervical range of motion.

Exclusion Criteria:

* None.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is based on 100 whiplash patients which underwent a measurment of the cervical movements and gave permission to recontact them for further research.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Active- and passive cervical range of motion measured with the 3Space InsideTrak HP system. | 31-12-2010

SECONDARY OUTCOMES:
Investigate the correlation between active- and passive cervical movement restraints and: NRS, TSK, PCS, NDI, CES-D, TAS, EPQ, CFQ, Holmes-Rahe scale, Rand 36, PSS-SR | 31-12-2010

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Patijn, dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands